CLINICAL TRIAL: NCT01905423
Title: Optimization of Mass Drug Administration With Existing Drug Regimens for Lymphatic Filariasis and Onchocerciasis
Acronym: DOLF-Indo
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gary Weil, MD, Professor of Medicine/ Microbiology, Washington University School of Medicine
Other Study IDs: 201103313
Record Dates: First submitted 2012-04-11; First posted 2013-07-23 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Lymphatic Filariasis; Soil Transmitted Helminth Infections
Keywords: Filariasis; Albendazole; Diethylcarbamazine; STH Soil Transmitted Helminths; MDA Mass Drug Administration
MeSH Terms: conditions — Elephantiasis, Filarial; Filariasis | interventions — Albendazole; Albumins; Diethylcarbamazine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Study procedures include collection of finger prick blood that will be tested for microfilaremia and for serology testing (antigenemia and antibody testing). We will also collect stool samples to detect STH infections.
  All assays will be performed in Indonesia (filarial serology tests, MF smears, stool examinations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Paga (annual MDA): This group includes eligible residents of the village of Paga. This cohort will receive once yearly MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Paga received a total of three rounds of MDA over a period of 24 months (once every 12 months).
  Interventions: Drug: Albendazole (annual); Drug: Diethylcarbamazine (annual)
- Lewomada (annual MDA): This group includes eligible residents of the village of Lewomada. This cohort will receive once yearly MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Lewomada received a total of three rounds of MDA over a period of 24 months (once every 12 months).
  Interventions: Drug: Albendazole (annual); Drug: Diethylcarbamazine (annual)
- Pruda (semiannual MDA): This group includes eligible residents of the village of Pruda. This cohort will receive twice yearly MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will also be administered by the Indonesian Ministry of Health.
  Pruda received a total of five rounds of MDA over a period of 24 months (once every 6 months).
  Interventions: Drug: Albendazole (semiannual); Drug: Diethylcarbamazine (semiannual)
- Pekalongan (annual MDA): This group includes the villages of Banyurip Ageng and Jenggot. This cohort will receive once yearly MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Pekalongan study sites were dropped after the first year follow-up due to lower than expected rates of lymphatic filariasis.
  Interventions: Drug: Albendazole (annual); Drug: Diethylcarbamazine (annual)
- Pekalongan (semiannual MDA): This group includes the villages of Kertoharjo and Pabean. This cohort will receive twice yearly MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will also be administered by the Indonesian Ministry of Health.
  Pekalongan study sites were dropped after the first year follow-up due to lower than expected rates of lymphatic filariasis.
  Interventions: Drug: Albendazole (semiannual); Drug: Diethylcarbamazine (semiannual)

INTERVENTIONS:
Drug: Albendazole (annual) — Albendazole 400 mg pnce annually
  Other Names: Albenza (Albendazole, also known as ALB)
  Groups: Lewomada (annual MDA); Paga (annual MDA); Pekalongan (annual MDA)
Drug: Diethylcarbamazine (annual) — Diethylcarbamazine 6 mg/kg once annually
  Other Names: Diethylcarbamazine, Also known as DEC, (N, N-diethyl-4-methyl-1-piperazine carboxamide dihydrogen citrate). ATC Code: P02CB02 QP52AH02
  Groups: Lewomada (annual MDA); Paga (annual MDA); Pekalongan (annual MDA)
Drug: Albendazole (semiannual) — Albendazole 400 mg twice annually
  Other Names: Albenza (Albendazole, also known as ALB)
  Groups: Pekalongan (semiannual MDA); Pruda (semiannual MDA)
Drug: Diethylcarbamazine (semiannual) — Diethylcarbamazine 6 mg/kg twice annually
  Other Names: Diethylcarbamazine, Also known as DEC, (N, N-diethyl-4-methyl-1-piperazine carboxamide dihydrogen citrate). ATC Code: P02CB02 QP52AH02
  Groups: Pekalongan (semiannual MDA); Pruda (semiannual MDA)

SUMMARY:
Approximately 3,500 people will participate per year. The study population will include females and males over 5 years of age who live in filariasis endemic areas. The study will be performed in Indonesia in B. timori and W. bancrofti endemic areas over a period of 4 years. Participants will be studied only once in cross-sectional surveys. Some subjects may be included in more than one annual population survey, but this is not a longitudinal study. Purpose of the study is to evaluate different mass drug administration (MDA) regimens for lymphatic filariasis and also to study the impact of MDA on soil transmitted helminth infections (STH). MDA will administered by others (e.g., Ministry of Health). Results of this study may enhance efforts to control and eliminate these important neglected tropical diseases.

The investigators will test the hypothesis that accelerated mass drug administration will be superior to annual MDA for elimination of lymphatic filariasis and for control of soil transmitted helminth infections (STH):

1. Compare the relative impact and cost effectiveness of annual vs. twice yearly mass drug administration (MDA) for elimination of lymphatic filariasis (LF).
2. Study the impact of annual vs. semiannual MDA on soil transmitted helminth (STH) infection in these populations.

DETAILED DESCRIPTION:
Lymphatic filariasis (LF) is a deforming and disabling infectious disease that causes elephantiasis and genital deformity (especially hydroceles). The infection affects some 120 million people in 81 countries in tropical and subtropical regions with well over 1 billion people at risk of acquiring the disease. LF is caused by Wuchereria bancrofti and Brugia spp. (B. malayi and B.timori), nematode parasites that are transmitted by mosquitoes. This study is based on the assumption that currently used mass drug administration (MDA) regimens and schedules are not optimal for achieving elimination of LF. These regimens (either annual Albendazole (Alb) 400 mg plus diethylcarbamazine (DEC) 6 mg/kg or Alb 400 mg plus ivermectin (Iver) 200 µg/kg for LF) were developed more than 10 years ago.

Drugs used for LF MDA are also active against soil transmitted helminth infections (STH, e.g., Ascaris, Hookworm, and Trichuris). De-worming campaigns using anthelminthics usually target special groups of the population, such as schoolchildren, and have limited impact on the transmission. Treatment of the total population and semiannual treatments may reduce re-infection considerably and will most likely lead to reduced infection densities and infection prevalences. Suppression of STH is an important ancillary benefit of MDA programs for filarial infections.

Purpose: The study aims to compare the effectiveness once yearly (1X) versus twice yearly (2X) mass drug administration (MDA) for the elimination of lymphatic filariasis and for control of soil-transmitted helminths (intestinal parasites) in large populations. Mass drug administration will be provided by the Indonesia Ministry of Health. This project will assess the impact of the public health program.

Procedures: Study procedures include collection of finger prick blood that will be tested for microfilaremia and for serology testing (antigenemia and antibody testing). Stool samples will be collected to detect STH infections. All assays will be performed in Indonesia (filarial serology tests, blood smears for detection of microfilariae (MF), and stool examinations for detection of worm eggs).

Washington University researchers developed the protocol, will provide training and guidance to Indonesian researchers, and work with them to analyze the data. Indonesian researchers will consent the participants, obtain stool and blood specimens, perform laboratory tests on the specimens, and enter data on participants and lab results.

ELIGIBILITY:
Inclusion Criteria:

* Areas should be endemic for filariasis and have limited or no prior experience with MDA. Males and Females greater than or equal to 5 years of age.

Exclusion Criteria:

* Children less than 5 years of age.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study populations are people who live in areas of Indonesia that are endemic for lymphatic filariasis.
Sampling Method: Non-Probability Sample
Enrollment: 17108 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter U Fischer, Ph.D., Principal Investigator — Washington University School of Medicine; Gary J Weil, MD, Principal Investigator — Washington University School of Medicine; Taniawati Supali, Ph.D., Study Director — Indonesia University
Locations (1):
- University of Indonesia, Department of Parasitology, Jakarta, Java, Indonesia

REFERENCES:
- See also: Death to Onchocerciasis and Lymphatic Filariasis (DOLF) — http://www.dolf.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cross-sectional study. The final end points of the study are measures of community prevalence. Participant involvement in the study ended after each survey period. Participants were not followed across survey periods, but could be and were likely recruited into more than one survey period.
Groups:
- Paga (1x Annual MDA): The village of Paga received once annual MDA for a total of 3 rounds over 24 months.
- Lewomada (1x Annual MDA): Village of Lewomada received once annual MDA for a total of 3 rounds over 24 months.
- Pruda (2x Annual MDA): The village of Pruda received twice annual MDA for a total of 5 rounds over 24 months.
- Pekalongan (1x Annual MDA): The Pekalongan study site was dropped from further analysis after the first year follow-up due to lower than expected prevalence of lymphatic filariasis infections. Baseline and year 1 follow-up results are presented separately from the other study sites. This group received one round of MDA and was surveyed one year later.
- Pekalongan (2x Annual MDA): The Pekalongan study site was dropped from further analysis after the first year follow-up due to lower than expected prevalence of lymphatic filariasis infections. Baseline and year 1 follow-up results are presented separately from the other study sites. This group received two rounds of MDA and was surveyed one year later.
Period: Overall Study
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Started | 4456 | 3297 | 4111 | 2757 | 2487
Baseline | 1443 | 722 | 1033 | 1482 | 1326
Year 1 Follow-up | 994 | 846 | 1007 | 1275 | 1161
Year 2 Follow-up | 1114 | 858 | 1043 | 0 | 0
Year 3 Follow-up | 905 | 871 | 1028 | 0 | 0
Completed | 4456 | 3297 | 4111 | 2757 | 2487
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Number of Baseline Participants that is reported is actually the total number of participants surveyed before the first round of treatment. This is a cross-sectional study. The Pekalongan study site was dropped from further study following the first year follow-up due to lower than expected prevalence of lymphatic filariasis infections.
Groups:
- Annual MDA Treated Group (Paga); Annual MDA Treated Group (Lewomada): This group will receive annual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Albendazole and diethylcarbamazine: Albendazole 400 mg plus diethylcarbamazine 6 mg/kg once yearly vs twice yearly
- Semiannual MDA Treated Group: This group will receive semiannual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will also be administered by the Indonesian Ministry of Health.
  Albendazole and diethylcarbamazine: Albendazole 400 mg plus diethylcarbamazine 6 mg/kg once yearly vs twice yearly
- Annual MDA Treated Group (Pekalongan): The Pekalongan study site was dropped from further analysis after the first year follow-up due to lower than expected prevalence of lymphatic filariasis infections. Baseline and year 1 follow-up results are presented separately from the other study sites.
  This group will receive annual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Albendazole and diethylcarbamazine: Albendazole 400 mg plus diethylcarbamazine 6 mg/kg once yearly vs twice yearly
- Semiannual MDA Treated Group (Pekalongan): The Pekalongan study site was dropped from further analysis after the first year follow-up due to lower than expected prevalence of lymphatic filariasis infections. Baseline and year 1 follow-up results are presented separately from the other study sites.
  This group will receive semiannual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will also be administered by the Indonesian Ministry of Health.
  Albendazole and diethylcarbamazine: Albendazole 400 mg plus diethylcarbamazine 6 mg/kg once yearly vs twice yearly
- Total: Total of all reporting groups
Arm/Group | Annual MDA Treated Group (Paga) | Annual MDA Treated Group (Lewomada) | Semiannual MDA Treated Group | Annual MDA Treated Group (Pekalongan) | Semiannual MDA Treated Group (Pekalongan) | Total
Number analyzed (Participants) | 1443 | 722 | 1033 | 1482 | 1326 | 6006
Age, Customized [Count of Participants; unit: Participants]
  Age at Baseline (pre-MDA): 15 years and younger | 597 | 285 | 374 | 353 | 372 | 1981
  Age at Baseline (pre-MDA): Older than 15 | 794 | 437 | 653 | 1129 | 954 | 3967
  Age at Baseline (pre-MDA): Age unknown | 52 | 0 | 6 | 0 | 0 | 58
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender at Baseline (pre-MDA): Females | 897 | 411 | 545 | 816 | 721 | 3390
  Gender at Baseline (pre-MDA): Males | 546 | 311 | 488 | 666 | 605 | 2616
  Gender at Baseline (pre-MDA): Gender unknown | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Microfilaria in Blood as Determined by Microscopy of Participant Blood
Description: Microfilariae (filarial parasites) will be detected in blood smears by microscopy. Samples will be collected in annual and semiannual community surveys. Prevalence rates (a measure of the disease rates in the population sampled) are expressed as % positive for microfilaremia (having microfilaria in the blood).
Time Frame: 3 years
Population: The Pekalongan study sites were dropped after the first year due to lower than expected prevalence of lymphatic filariasis infections. The overall number of participants analyzed for each group may be slightly less than the total sample size for that group due to the fact that not all data was collected for all participants.
Measure: Count of Participants; unit: Participants
Groups:
- Paga (1x Annual MDA); Lewomada (1x Annual MDA); Pekalongan (1x Annual MDA); Pekalongan (2x Annual MDA): Participants from this village receive annual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Albendazole and diethylcarbamazine Annual: Albendazole and diethylcarbamazine Annual Albendazole 400 mg plus diethylcarbamazine 6 mg/kg once yearly
- Pruda (2x Annual MDA): Participants from this village receive semiannual MDA (Albendazole 400 mg plus diethylcarbamazine 6 mg/kg) which will also be administered by the Indonesian Ministry of Health.
  Albendazole and diethylcarbamazine Semiannual: Albendazole and diethylcarbamazine Semiannual Albendazole 400 mg plus diethylcarbamazine 6 mg/kg twice yearly
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 4401 | 3297 | 4079 | 2730 | 2427
Participants
  Baseline (pre-MDA): number analyzed (Participants) | 1391 | 722 | 1027 | 1455 | 1266
  Baseline (pre-MDA) | 54 | 36 | 146 | 46 | 45
  Year 1: number analyzed (Participants) | 994 | 846 | 982 | 1275 | 1161
  Year 1 | 11 | 9 | 37 | 28 | 30
  Year 2: number analyzed (Participants) | 1114 | 858 | 1043 | 0 | 0
  Year 2 | 6 | 6 | 15 | 0 | 0
  Year 3: number analyzed (Participants) | 902 | 871 | 1027 | 0 | 0
  Year 3 | 0 | 3 | 12 | 0 | 0

2. Secondary Outcome: Prevalence of Positive Brugia Rapid Antifilarial Antibody Tests
Description: This outcome is reported as the frequency of participants with positive Brugia Rapid antifilarial antibody tests. Data was only collected at baseline and at year 3 for this outcome measure and no antibody data was collected for the Pekalongan study sites.
Time Frame: 3 years
Population: This outcome data was only collected at baseline and at year 3 for Paga & Pruda and no antibody data was collected at all for the Pekalongan study sites. The overall number of participants analyzed for each group may be less than the total sample size for that group due to the fact that not all data was collected for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 2308 | 3297 | 2054 | 0 | 0
Participants
  Baseline: number analyzed (Participants) | 1403 | 722 | 1027 | 0 | 0
  Baseline | 175 | 229 | 297 | 0 | 0
  Year 1: number analyzed (Participants) | 0 | 846 | 0 | 0 | 0
  Year 1 | 0 | 168 | 0 | 0 | 0
  Year 2: number analyzed (Participants) | 0 | 858 | 0 | 0 | 0
  Year 2 | 0 | 134 | 0 | 0 | 0
  Year 3: number analyzed (Participants) | 905 | 871 | 1027 | 0 | 0
  Year 3 | 16 | 36 | 37 | 0 | 0

3. Secondary Outcome: Prevalence of Circulating Filarial Antigen in Blood as Determined by ICT Card Test
Description: Prevalence of filarial antigenemia (detected with the Binax Filariasis Now card test "ICT" card test) among the population surveyed. Prevalence data are expressed as %.
Time Frame: 3 years
Population: This outcome data was not collected for Paga at year 3 or for Pekalongan sites after year 1 (Pekalongan study site was dropped completely after year 1). The overall number of participants analyzed for each group may be less than the total sample size for that group due to the fact that not all data was collected for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 3511 | 3297 | 4095 | 2696 | 2407
Participants
  Baseline: number analyzed (Participants) | 1403 | 722 | 1027 | 1448 | 1285
  Baseline | 14 | 47 | 235 | 118 | 102
  Year 1: number analyzed (Participants) | 994 | 846 | 998 | 1248 | 1122
  Year 1 | 0 | 12 | 91 | 51 | 63
  Year 2: number analyzed (Participants) | 1114 | 858 | 1043 | 0 | 0
  Year 2 | 2 | 13 | 106 | 0 | 0
  Year 3: number analyzed (Participants) | 0 | 871 | 1027 | 0 | 0
  Year 3 | 0 | 36 | 72 | 0 | 0

4. Secondary Outcome: Prevalence of Ascaris Infection
Description: Prevalence of Ascaris infection is defined by the number of participants with any Ascaris worm eggs present in their stool sample as analyzed with microscopy.
Time Frame: 2 Years
Population: The Pekalongan study sites were dropped after the first year. No soil transmitted helminth infection data was collected after year 2. The overall number of participants analyzed for each group may be slightly less than the total sample size for that group due to the fact that not all data was collected for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 708 | 1230 | 523 | 699 | 792
Participants
  Baseline: number analyzed (Participants) | 147 | 375 | 132 | 474 | 618
  Baseline | 88 | 56 | 34 | 19 | 58
  Year 1: number analyzed (Participants) | 317 | 357 | 202 | 225 | 174
  Year 1 | 135 | 17 | 7 | 11 | 6
  Year 2: number analyzed (Participants) | 244 | 498 | 189 | 0 | 0
  Year 2 | 107 | 18 | 3 | 0 | 0

5. Secondary Outcome: Prevalence of Hookworm Infection
Description: Prevalence of hookworm infection is defined by the number of participants with any hookworm eggs present in their stool sample as analyzed with microscopy.
Time Frame: 2 years
Population: Hookworm prevalence was not analyzed for Pekalongan sites. Hookworm data was not collected after year 2 for any sites. The overall number of participants analyzed for each group may be slightly less than the total sample size for that group due to the fact that not all data was collected for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 708 | 1230 | 523 | 0 | 0
Participants
  Baseline: number analyzed (Participants) | 147 | 375 | 132 | 0 | 0
  Baseline | 25 | 226 | 35 | 0 | 0
  Year 1: number analyzed (Participants) | 317 | 357 | 202 | 0 | 0
  Year 1 | 118 | 118 | 90 | 0 | 0
  Year 2: number analyzed (Participants) | 244 | 498 | 189 | 0 | 0
  Year 2 | 65 | 97 | 87 | 0 | 0

6. Secondary Outcome: Prevalence of Trichuris Infection
Description: Prevalence of trichuris infection is defined by the number of participants with any trichuris worm eggs present in their stool sample as analyzed with microscopy.
Time Frame: 2 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Paga (1x Annual MDA) | Lewomada (1x Annual MDA) | Pruda (2x Annual MDA) | Pekalongan (1x Annual MDA) | Pekalongan (2x Annual MDA)
Number analyzed (Participants) | 708 | 1230 | 523 | 699 | 792
Participants
  Baseline: number analyzed (Participants) | 147 | 375 | 132 | 474 | 618
  Baseline | 68 | 45 | 8 | 120 | 352
  Year 1: number analyzed (Participants) | 317 | 357 | 202 | 225 | 174
  Year 1 | 93 | 25 | 8 | 35 | 65
  Year 2: number analyzed (Participants) | 244 | 498 | 189 | 0 | 0
  Year 2 | 84 | 23 | 13 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will be monitored for adverse events related to blood collection at each year of observation.
Description: This is a minimal risk and nonintervention study. Adverse events are not expected to be an issue. However, subjects will be monitored for adverse events related to blood collection.
Groups:
- Paga (Annual MDA): This group includes eligible residents of the village of Paga. This cohort will receive once yearly MDA (albendazole 400 mg + diethylcarbamazing 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Paga received a total of three rounds of MDA over a period of 24 months (once every 12 months).
- Lewomada (Annual MDA): This group includes eligible residents of the village of Lewomada. This cohort will receive once yearly MDA (albendazole 400 mg + diethylcarbamazing 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Lewomada received a total of three rounds of MDA over a period of 24 months (once every 12 months).
- Pruda (Semiannual MDA): This group includes eligible residents of the village of Pruda. This cohort will receive twice yearly MDA (albendazole 400 mg + diethylcarbamazing 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Pruda received a total of five rounds of MDA over a period of 24 months (once every 6 months).
- Pekalongan (Annual MDA): This group includes villages of Banyurip Ageng and Jenggot. This cohort will receive once yearly MDA (albendazole 400 mg + diethylcarbamazing 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Pekalongan study sites were dropped after the first year follow-up due to lower than expected rates of lymphatic filariasis.
- Pekalongan (Semiannual MDA): This group includes villages of Kertoharjo and Pabean. This cohort will receive twice yearly MDA (albendazole 400 mg + diethylcarbamazing 6 mg/kg) which will be administered by the Indonesian Ministry of Health as part of their national filariasis elimination program.
  Pekalongan study sites were dropped after the first year follow-up due to lower than expected rates of lymphatic filariasis.
Arm/Group | Paga (Annual MDA) | Lewomada (Annual MDA) | Pruda (Semiannual MDA) | Pekalongan (Annual MDA) | Pekalongan (Semiannual MDA)
All-Cause Mortality (participants affected / at risk) | 0/4456 | 0/3297 | 0/4111 | 0/2757 | 0/2487
Serious Adverse Events (participants affected / at risk) | 0/4456 | 0/3297 | 0/4111 | 0/2757 | 0/2487
Other Adverse Events (participants affected / at risk) | 0/4456 | 0/3297 | 0/4111 | 0/2757 | 0/2487

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT01905423/Prot_SAP_000.pdf